CLINICAL TRIAL: NCT06541132
Title: Positive Association Between Ultrasonographic Fatty Liver Indicator and the Severity of Coronary Artery Disease
Brief Title: Positive Association of US-FLI With the Severity of CAD
Status: Recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Tingqiu Wang, Principal Investigator, Chongqing Medical University
Other Study IDs: ChongqingM
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease of Significant Bypass Graft; Metabolic Dysfunction-associated Fatty Liver Disease; SYNTAX Score; Ultrasonography
Keywords: Coronary Artery Disease; Metabolic Dysfunction-associated Fatty Liver Disease; SYNTAX score; Ultrasonography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-CAD group: non-coronary artery disease group
- CAD group: coronary artery disease group
  Interventions: Other: Observational study without human intervention
- SS≤22 group: SYNTAX score ≤22
- SS≥23 group: SYNTAX score ≥23
  Interventions: Other: Observational study without human intervention

INTERVENTIONS:
Other: Observational study without human intervention — Observational study without human intervention
  Groups: CAD group; SS≥23 group

SUMMARY:
As a multisystem disease, metabolic dysfunction-associated fatty liver disease (MAFLD) is closely linked to the onset and progression of coronary heart disease (CHD). Ultrasonographic fatty liver indicator (US-FLI) is a semi-quantitative tool for evaluating the degree of hepatic steatosis. Our study aims to explore the relationship between US-FLI based on MAFLD and the severity of CHD.

DETAILED DESCRIPTION:
204 patients who had invasive coronary angiography performed between July 2022 and December 2023 at the cardiology department of the Second Affiliated Hospital of Chongqing Medical University were included in this study. Collect clinical information and abdominal ultrasound images from each patient. Hepatic steatosis which quantified by US-FLI was evaluated by the echo contrast between liver and kidney, posterior attenuation of ultrasound beam, areas of focal sparing, display of hepatic vessels, gallbladder wall and diaphragm. Fatty liver was diagnosed when US-FLI≥2. The severity of CHD was evaluated using the SYNTAX score (SS), and a total of 100 CHD patients were ultimately diagnosed. CHD patients were further divided into the low-risk group (SS ≤ 22) (54 cases) and the medium-high-risk group (SS≥23) (46 cases). Multivariate logistic regression model was used to assess the relationship between US-FLI and SS in patients with MAFLD. The receiver operating characteristic curve was used to determine the accuracy, sensitivity and specificity of US-FLI in predicting SS.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients underwent ICA due to chest pain, chest tightness or other reasons in our hospital from August 2022 to December 2023 were included in our study

Exclusion Criteria:

* Incomplete clinical data
* previous coronary stent implantation
* no abdominal ultrasound examination
* poor ultrasound image quality
* congenital heart disease
* tumor
* thyroid diseases and infectious diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All research subjects were from the Second Affiliated Hospital of Chongqing Medical University
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
SYNTAX score | at baseline
  The complexity of coronary artery disease (CAD) is a predictor of cardiovascular events in patients with >50 % diameter stenosis as determined by SYNTAX score. The range of US-FLI is 0-8. Fatty liver was diagnosed when US-FLI ≥ 2.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004
- [Background] Ballestri S, Nascimbeni F, Baldelli E, Marrazzo A, Romagnoli D, Targher G, Lonardo A. Ultrasonographic fatty liver indicator detects mild steatosis and correlates with metabolic/histological parameters in various liver diseases. Metabolism. 2017 Jul;72:57-65. doi: 10.1016/j.metabol.2017.04.003. Epub 2017 Apr 13. PMID 28641784
- [Background] Buckley AJ, Thomas EL, Lessan N, Trovato FM, Trovato GM, Taylor-Robinson SD. Non-alcoholic fatty liver disease: Relationship with cardiovascular risk markers and clinical endpoints. Diabetes Res Clin Pract. 2018 Oct;144:144-152. doi: 10.1016/j.diabres.2018.08.011. Epub 2018 Aug 28. PMID 30170074
- [Background] Liu Z, Que S, Xu J, Peng T. Alanine aminotransferase-old biomarker and new concept: a review. Int J Med Sci. 2014 Jun 26;11(9):925-35. doi: 10.7150/ijms.8951. eCollection 2014. PMID 25013373